CLINICAL TRIAL: NCT05164939
Title: Precision Medicine Intervention in Severe Asthma (PRISM) Study: Molecular Phenotyping of Participants With Severe Asthma to Determine Response to Biologic Therapies and Stability
Brief Title: Precision Medicine Intervention in Severe Asthma (PRISM) Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, Tae-Bum Kim, Professor, Asan Medical Center
Other Study IDs: 2019-1676
Record Dates: First submitted 2021-11-01; First posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-12

CONDITIONS: Severe Asthma
Keywords: biologics, multi-omics analysis
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, urine, exhaled breath, sputum, nasal epithelial cells, bronchial epithelial cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Korea-UK Precision Medicine Intervention in Severe Asthma (PRISM) study aims to identify molecular phenotypes of severe asthma by analyzing multi-omics data including genomics, epigenomics, transcriptomics, proteomics, metagenomics, and metabolomics.

DETAILED DESCRIPTION:
This is a prospective, observational cohort study. The participants are composed of the patients having severe asthma treated with biologic agents or conventional medication. Once enrolled, regular evaluation of clinical characteristics and obtainment of samples for omics analysis is conducted to identify clinically relevance molecular signals in severe asthmatics.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subject aged between 18 years and 80 years
* Give written informed consent prior to participation in the study including all procedures
* Comply with study protocol requirements
* Able to read, comprehend, and write at a sufficient level to complete study related materials
* Able to complete the study and all measurements
* All patients have been through a severe asthma protocol that have ascertained the diagnosis of severe asthma, maximised treatments and ensured adherence to therapy.
* Stable asthma therapy for at least a month before screening

Exclusion Criteria:

* As a result of medical interview, physical examination or screening investigation the investigators consider the subject unfit either because of risk to the subject due to the study or the influence this may have on the study results.
* A history of recreational drug use or allergy which in the opinion of the investigators contraindicates their participation.
* Participation within 3 months in any a trial testing a new molecular entity or drug.
* Those, in the opinion of the investigator, who may prove non-compliant with study procedures.
* Within 4 weeks of screening visit been hospitalized or required high dose oral corticosteroid (>30 mg prednisolone per day) therapy, asthma not been stable.
* Patients who have had prior treatment with bronchial thermoplasty, defined as completion of all thermoplasty treatment sessions within 6 months of screening
* History of significant pulmonary disease other than severe asthma.
* History of pulmonary eosinophilic syndrome or hyper eosinophilic syndrome.
* History of bronchopulmonary aspergillosis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with severe asthma
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Asthma exacerbations | baseline, 1month, 6month, 10 month
  Changes of number of asthma exacerbations

SECONDARY OUTCOMES:
Asthma symptom control | baseline, 1month, 6month, 10 month
  Changes in symptom score using the Asthma Control Test (ACT)
Quality of Life Questionnaire | baseline, 1month, 6month, 10 month
  Change in quality of life using EuroQol-5 dimension
Rhinosinusitis symptoms | baseline, 1month, 6month, 10 month
  Change in nasal symptoms using 22-item Sino-Nasal Outcome Test (SNOT-22)
Forced Exahled Volume in 1 second (FEV1) | baseline, 1month, 6month, 10 month
  Changes in FEV1 in liter and % from baseline
Forced Vital Capacity (FVC) | baseline, 1month, 6month, 10 month
  Changes in FVC in liter and % from baseline
Fraction of exhaled nitric oxide, FENO | baseline, 1month, 6month, 10 month
  Changes in FENO in ppb
Induced sputum eosinophil | baseline, 1month, 6month, 10 month
  Changes in sputum eosinophil
Blood eosinophils | baseline, 1month, 6month, 10 month
  Changes in blood eosinophil

CONTACTS AND LOCATIONS:
Overall Officials: Tae-Bum Kim, Principal Investigator — Asan Medical Center; Kian Fan Chung, Principal Investigator — Imperial College London
Locations (2):
- Asan medical center, Seoul, Songpagu, South Korea
- Imperial college, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
undecided

REFERENCES:
- [Derived] Lee Y, Kim H, Lee CE, Lee BJ, Kim MH, Park SY, Kim BK, Kim SH, Kim SH, Park HK, Lee T, Shim JS, Park CS, Park HK, Kwon JW, Kim S, Nam YH, Yang MS, Jung JW, Kim TB. Siglec-8 as a Biomarker for Predicting Anti-IL-5 Response in Severe Asthma. Allergy Asthma Immunol Res. 2025 Nov;17(6):742-753. doi: 10.4168/aair.2025.17.6.742. PMID 41330705
- [Derived] Kang YR, Kim H, Lee CE, Jung JW, Moon JY, Park SY, Kim SH, Yang MS, Kim BK, Kwon JW, Park HK, Nam YH, Cho YJ, Lee T, Adcock IM, Bhavsar P, Chung KF, Kim TB. Serum and urine eosinophil-derived neurotoxin (EDN) levels predict biologic response in severe asthma. World Allergy Organ J. 2025 Jan 9;18(1):100990. doi: 10.1016/j.waojou.2024.100990. eCollection 2025 Jan. PMID 39896201
- [Derived] Park K, Lee JH, Shin E, Jang HY, Song WJ, Kwon HS, Cho YS, Lee JE, Adcock I, Chung KF, Lee JS, Won S, Kim TB. Single-cell RNA sequencing reveals transcriptional changes in circulating immune cells from patients with severe asthma induced by biologics. Exp Mol Med. 2024 Dec;56(12):2755-2762. doi: 10.1038/s12276-024-01368-y. Epub 2024 Dec 13. PMID 39672815
- [Derived] Pham DD, Lee JH, Kwon HS, Song WJ, Cho YS, Kim H, Kwon JW, Park SY, Kim S, Hur GY, Kim BK, Nam YH, Yang MS, Kim MY, Kim SH, Lee BJ, Lee T, Park SY, Kim MH, Cho YJ, Park C, Jung JW, Park HK, Kim JH, Moon JY, Adcock I, Bhavsar P, Chung KF, Kim TB. Prospective direct comparison of biologic treatments for severe eosinophilic asthma: Findings from the PRISM study. Ann Allergy Asthma Immunol. 2024 Apr;132(4):457-462.e2. doi: 10.1016/j.anai.2023.11.005. Epub 2023 Nov 17. PMID 37977324